CLINICAL TRIAL: NCT02240498
Title: A Phase 1 Study to Assess Safety and Feasibility of Methylene Blue Photodynamic Therapy to Sterilize Deep Tissue Abscess Cavities
Brief Title: Safety and Feasibility Study of Methylene Blue Photodynamic Therapy to Sterilize Deep Tissue Abscess Cavities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Timothy Baran, Assistant Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00049677
Record Dates: First submitted 2014-09-03; First posted 2014-09-15 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Abscess
Keywords: Abscess; Drainage
MeSH Terms: conditions — Abscess | interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- MB-PDT, 5 min illumination (Experimental): Each subject in this group will receive methylene blue, 20% I.V. fat emulsion, insertion of optical fiber, and laser illumination, 5 minutes.
  Interventions: Drug: Methylene Blue; Drug: 20% I.V. Fat Emulsion; Device: Insertion of optical fiber; Device: Laser illumination, 5 minutes
- MB-PDT, 10 min illumination (Experimental): Each subject in this group will receive methylene blue, 20% I.V. fat emulsion, insertion of optical fiber, optical spectroscopy measurement, and laser illumination, 10 minutes.
  Interventions: Drug: Methylene Blue; Drug: 20% I.V. Fat Emulsion; Device: Insertion of optical fiber; Device: Laser illumination, 10 minutes; Device: Optical spectroscopy measurement
- MB-PDT, 15 min illumination (Experimental): Each subject in this group will receive methylene blue, 20% I.V. fat emulsion, insertion of optical fiber, optical spectroscopy measurement, and laser illumination, 15 minutes.
  Interventions: Drug: Methylene Blue; Drug: 20% I.V. Fat Emulsion; Device: Insertion of optical fiber; Device: Laser illumination, 15 minutes; Device: Optical spectroscopy measurement
- MB-PDT, 20 min illumination (Experimental): Each subject in this group will receive methylene blue, 20% I.V. fat emulsion, insertion of optical fiber, optical spectroscopy measurement, and laser illumination, 20 minutes.
  Interventions: Drug: Methylene Blue; Drug: 20% I.V. Fat Emulsion; Device: Insertion of optical fiber; Device: Laser illumination, 20 minutes; Device: Optical spectroscopy measurement
- MB-PDT, 25 min illumination (Experimental): Each subject in this group will receive methylene blue, 20% I.V. fat emulsion, insertion of optical fiber, optical spectroscopy measurement, and laser illumination, 25 minutes.
  Interventions: Drug: Methylene Blue; Drug: 20% I.V. Fat Emulsion; Device: Insertion of optical fiber; Device: Laser illumination, 25 minutes; Device: Optical spectroscopy measurement
- MB-PDT, 30 min illumination (Experimental): Each subject in this group will receive methylene blue, 20% I.V. fat emulsion, insertion of optical fiber, optical spectroscopy measurement, and laser illumination, 30 minutes.
  Interventions: Drug: Methylene Blue; Drug: 20% I.V. Fat Emulsion; Device: Insertion of optical fiber; Device: Laser illumination, 30 minutes; Device: Optical spectroscopy measurement

INTERVENTIONS:
Drug: Methylene Blue — Administration of 1 mg/mL methylene blue to the abscess cavity, followed by a 10 minute incubation interval. After this incubation interval, the methylene blue solution will be aspirated from the cavity and flushed twice with sterile saline.
  Other Names: Methylene Blue Injection, USP 1%
Drug: 20% I.V. Fat Emulsion — The abscess cavity will be filled with sterile 1% Intralipid solution to gently distend the cavity and, through efficient light scattering, to homogenize the light dose to the walls of the cavity. After laser illumination, the Intralipid will be aspirated from the cavity.
  Other Names: Intralipid 20%
Device: Insertion of optical fiber — A sterile, FDA-approved optical fiber will be advanced to the approximate center of the abscess cavity via the drainage catheter under image guidance. Following laser illumination, the fiber will be withdrawn.
  Other Names: Vascular Solutions VariLase Bright Tip Fiber M7106
Device: Laser illumination, 5 minutes — Laser illumination will be delivered via the optical fiber for a duration of 5 minutes. The fluence rate will be set such that the maximum fluence rate at the abscess wall is 20 mW/cm2.
  Other Names: Modulight ML7710-PDT Laser System
  Arms: MB-PDT, 5 min illumination
Device: Laser illumination, 10 minutes — Laser illumination will be delivered via the optical fiber for a duration of 10 minutes. The fluence rate will be set such that the maximum fluence rate at the abscess wall is 20 mW/cm2.
  Other Names: Modulight ML7710-PDT Laser System
  Arms: MB-PDT, 10 min illumination
Device: Laser illumination, 15 minutes — Laser illumination will be delivered via the optical fiber for a duration of 15 minutes. The fluence rate will be set such that the maximum fluence rate at the abscess wall is 20 mW/cm2.
  Other Names: Modulight ML7710-PDT Laser System
  Arms: MB-PDT, 15 min illumination
Device: Laser illumination, 20 minutes — Laser illumination will be delivered via the optical fiber for a duration of 20 minutes. The fluence rate will be set such that the maximum fluence rate at the abscess wall is 20 mW/cm2.
  Other Names: Modulight ML7710-PDT Laser System
  Arms: MB-PDT, 20 min illumination
Device: Laser illumination, 25 minutes — Laser illumination will be delivered via the optical fiber for a duration of 25 minutes. The fluence rate will be set such that the maximum fluence rate at the abscess wall is 20 mW/cm2.
  Other Names: Modulight ML7710-PDT Laser System
  Arms: MB-PDT, 25 min illumination
Device: Laser illumination, 30 minutes — Laser illumination will be delivered via the optical fiber for a duration of 30 minutes. The fluence rate will be set such that the maximum fluence rate at the abscess wall is 20 mW/cm2.
  Other Names: Modulight ML7710-PDT Laser System
  Arms: MB-PDT, 30 min illumination
Device: Optical spectroscopy measurement — A fiber-optic probe that has undergone high-level disinfection will be advanced through the drainage catheter/needle in order to make gentle contact with the wall of the cavity. Low-intensity white light will be delivered by a tungsten halogen lamp by a single fiber within the probe, and detected by eight other fibers within the probe. Following this, low-power laser light will be delivered by a fiber-coupled laser diode at 640 nm in order to excite methylene blue fluorescence. Emitted fluorescence will similarly be collected by the eight detection fibers contained within the probe. Upon completion of these measurements, the fiber-optic probe will be withdrawn, gently wiped with sterile gauze, and returned to the procedure cart.
  Arms: MB-PDT, 10 min illumination; MB-PDT, 15 min illumination; MB-PDT, 20 min illumination; MB-PDT, 25 min illumination; MB-PDT, 30 min illumination

SUMMARY:
The objectives of this Phase 1 study are to evaluate the safety and feasibility of methylene-blue-mediated photodynamic therapy (MB-PDT) performed at the time of abscess drainage to treat deep tissue abscesses. Safety will be evaluated by physical examination and imaging and laboratory studies in order to identify adverse events that may be induced by MB-PDT. We hypothesize that MB-PDT will be a safe and feasible intervention for this patient population. Optical measurements will additionally be performed at the abscess wall to determine optical properties and methylene blue uptake.

DETAILED DESCRIPTION:
Deep tissue abscesses remain a significant cause of morbidity, mortality, and hospital stay despite improved surgical techniques and increasing use of perioperative antibiotics. Mortality ranges from 80-100% in undrained collections and, in patients with intraperitoneal abscesses, reported hospital stays have been 21-47 days. The development of image-guided percutaneous drainage accompanied by antimicrobial treatment has been shown to improve patient outcomes and can significantly reduce mortality in uncomplicated fluid collections to 5% and morbidity to 10-15%. Even under favorable conditions, the use of long-term antibiotics increases the risk of acquired resistance and incidence of polymicrobial infection, which may limit future options for antibiotic treatment. Further, in 23% of patients, percutaneous drainage and intravenous antibiotics fail, requiring open surgical drainage, particularly in patients with abscesses infected with yeast or abscesses due to a pancreatic process.

Photodynamic therapy (PDT), which exerts antimicrobial activity through the generation of reactive oxygen species, may serve as a useful adjunct to current standard care of treating deep tissue abscesses by reducing the microbial burden following drainage. Recent work from our group demonstrated the effectiveness of methylene blue photodynamic therapy (MB-PDT) against organisms within primary aspirate fluid obtained from 32 patients who underwent image-guided percutaneous drainage of an abscess cavity. We found that MB-PDT was effective against multiple classes of organisms, including yeast and those displaying drug resistance. In these complex samples, we found no evidence of resistance to MB-PDT. These preclinical results obtained with samples harvested from the kinds of abscesses that we propose to treat provide a compelling rationale for evaluating the technical feasibility and safety of advancing optical fibers through catheters into an abscess cavity and performing PDT at the time of drainage. This clinical strategy would offer a wide range of potential health benefits to patients with deep tissue abscess. Among these advantages are reduced surgical intervention, decreased spread of infection, shortened course of post-treatment antibiotic therapy, and decreased selective pressure for antibiotic resistance. Ultimately, this would promote early recovery, shorten hospital stay, and lead to lower overall health care costs for patients undergoing image-guided percutaneous abscess drainage.

Image guided percutaneous drainage is performed at the University of Rochester using CT, ultrasound, or fluoroscopy. Focused imaging is performed, which confirms that the collection is amenable to drainage. The site is prepared and draped in the usual sterile fashion. The overlying skin is anesthetized with 1% lidocaine. A Hawkins/micropuncture needle is inserted, and the location confirmed under image guidance. The needle is advanced and placement within the collection is confirmed with imaging. Syringe aspiration of the abscess material is collected and sent for gram stain and culture. The needle is exchanged for a dilator and the 018 wire is replaced with a Coon's wire. If abscess collection contains multiple loculations, the end of the Coon's wire will be used to break up the loculations. The tract is further dilated with a transitional dilator followed by placement of an appropriate sized All Purpose Draining Locking pigtail catheter (8-14 French) into the fluid collection. The abscess will be drained by aspiration with a syringe. The catheter will be secured to the skin using 2-0 silk or stat-lock, dressed appropriately and connected to a drainage bag.

After drainage, the cavity will be flushed with sterile saline as per routine procedure. A fiber-optic probe that has undergone high-level disinfection will be advanced through the same catheter/needle in order to make gentle contact with the wall of the cavity. Low-intensity white light will be delivered by a tungsten halogen lamp by a single fiber within the probe, and detected by eight other fibers within the probe. Following this, low-power laser light will be delivered by a fiber-coupled laser diode in order to excite methylene blue fluorescence. Emitted fluorescence will similarly be collected by the eight detection fibers contained within the probe. Upon completion of these measurements, the fiber-optic probe will be withdrawn, gently wiped with sterile gauze, and returned to the procedure cart. The total time required for both reflectance and fluorescence measurements generally ranges from 10-60 seconds.

Following this, and using the same catheter, the cavity will then be filled with sterile, clinical grade methylene blue solution diluted 10-fold from its stock concentration of 10 mg/mL. The volume introduced will be matched to the cavity volume, which we estimate will not exceed 270 mL. In the unlikely case of the entire methylene blue dose escaping into systemic circulation, this results in a full body dose of 3.85 mg/kg for a typical patient weight of 70 kg. This is below the range for which adverse events have been reported for methylene blue.

After a 10-minute incubation interval, the methylene blue solution will be aspirated from the cavity and flushed twice with sterile saline. Optical measurements will then be repeated, as described above. Following this, the optical probe will be gently wiped with sterile gauze and sealed in a plastic bag for future high-level disinfection. Including the time required for positioning and capturing pre- and post-MB measurements, these optical measurements are expected to add less than four minutes to the overall procedure time.

The cavity will then be filled with sterile 1% Intralipid solution to gently distend the cavity and, through efficient light scattering, to homogenize the light dose to the walls of the cavity.

A sterile, FDA-approved optical fiber will be advanced to the approximate center of the abscess cavity via the same catheter under image guidance. The proximal end of the fiber is coupled to the output of a diode laser system emitting light at 665 nm, where methylene blue is activated optimally. Laser power will be delivered to the cavity at a constant fluence rate at the wall of 10 - 20 milliWatts (mW) cm-2. The laser power required to obtain the desired fluence rate at the wall will be calculated and documented on a written form in the procedure room based on the abscess size, with total laser power in the range of 1-2 W. The diode laser system being used is capable of measuring optical power, and will be used to directly measure the output from the optical fiber before treating each patient. These fluence rates are within an appropriate range for effective photodynamic therapy but well below the intensity at which modest thermal effects are observed in tissue. Immediately after laser irradiation, the Intralipid solution will be aspirated and the cavity again flushed with sterile saline.

Fluence escalation will be accomplished by systematically incrementing the duration of laser exposure according to a "3 + 3" dose escalation scheme. Under this design, the first three patients will receive a 5 minute exposure of laser light. If no dose-limiting toxicities are encountered, the exposure duration will be increased by 5 minutes in the next group of three patients. If one dose-limiting toxicity is encountered, the next group of patients will receive the same exposure duration as the previous group. If two or more dose-limiting toxicities are encountered, the exposure will be de-escalated by 5 minutes. This process will continue until the maximum number of patients are treated, or 6 patients are treated at a de-escalated dose. In order to avoid excessive increases in procedure duration, the maximum duration of laser exposure will be 30 minutes. A dose-limiting toxicity is defined as diminished clinical condition, with evidence of one or more of the following: (i) evidence of fat embolism; (ii) methylene blue escape during procedure with evidence of adverse reaction; (iii) imaging evidence of clinically significant, therapy-induced disruption of the abscess wall and damage to surrounding tissue.

Antibiotics as prescribed by the subject's primary team will be administered before the procedure and continued post-procedure. These are selected to ensure adequate coverage and taking into account subject allergies. Such administration is considered the standard of care, and serves to reduce the rate of post-procedure sepsis. The subject will also be administered intravenous antiemetics as needed prior to the procedure for nausea.

Following the procedure and as per routine care, a combination of IV and PO antibiotics will be continued to reduce the rate of post procedure sepsis. Antiemetics will also be continued as needed to reduce symptoms of nausea and vomiting. Narcotics will be prescribed and administered to control pain symptoms.

If the subject is an inpatient at the time of drainage, he/she will remain hospitalized post-procedure. If the subject is an outpatient at the time of drainage, he/she will be admitted to the hospital post-procedure only if clinically warranted. The study doctor or his designate will visit hospitalized subjects daily to assess progress and AEs. The subject's clinical course will be discussed daily with the primary clinical team. Hospitalized subjects will be discharged based upon response to drainage and clinical course only if clinical indicators (white blood cell count, heart rate, blood pressure, and temperature) are stable. If the subject remains hospitalized as a result of underlying health issues that are unrelated to study participation, the study doctor or his designate will continue daily visits through day 5 post-procedure, hospital discharge or until the drain is removed, whichever comes first. The PI will follow up with all non-hospitalized subjects daily by telephone through 7 days post-procedure.

All subjects will be seen again at one week following the procedure to further assess for progress, AEs and abscess resolution. As per departmental protocols and procedures, if the abscess has resolved at day 7 as evidenced by catheter output of less than 20 cc daily and limited imaging of the abscess cavity, the drainage catheter will be removed. If the abscess persists beyond 7 days despite drainage, the catheter will remain in place and be evaluated again at day 14. If the abscess persists at day 7 and if clinically indicated, additional procedures (i.e. repeat draining with a larger diameter catheter) will be performed. MB-PDT will not be repeated. Abscess resolution will be determined by either ultrasound or CT scan as outlined below. Imaging at the time of catheter removal is considered standard of care.

A study visit at day 7 post procedure is required of all subjects. If the catheter is left in at that time, a second visit will be required at day 14. If the catheter is removed at day 7 and there are no unresolved AEs, subject study participation will end after that visit. If any subject cannot return as has been scheduled, the visit will be rescheduled to their convenience. The visits at 7 and, if necessary, 14 days post procedure are primarily to determine the timing for catheter removal and are standard of care following percutaneous drainage.

At a minimum, CBC w/ diff and serum creatinine will be acquired prior to the procedure. Blood cultures will be obtained as clinically indicated, and drainage cultures will be obtained at day 0. Additional laboratory and imaging studies will be performed as deemed clinically necessary.

There is very minimal risk of systemic skin photosensitivity after exposure to methylene blue. Based on studies of the pharmacokinetics of methylene blue, it was found that the majority was rapidly converted to leucomethylene blue, which is photodynamically inactive. In clinical studies of MB-PDT with MB administered intratumorally, intravesically, and via gargling, no skin photosensitivity was reported. Subjects will be monitored for any evidence of skin photosensitivity reaction after the procedure. Due to the rapid conversion of MB to leucomethylene blue in systemic circulation and the lack of photosensitivity in previous studies, no special precautions will be taken to limit the exposure of subjects to light after the procedure.

The 21 subjects enrolled in the study will be followed until all clinical findings post image-guided drainage and MB-PDT have cleared. Each subject will be evaluated by imaging and laboratory studies at scheduled visits 7 days post procedure and, if necessary, 14 days post procedure. It is estimated that this study will take approximately 2 years to complete.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* If female, patient must have negative pregnancy test
* All patients with clinical symptoms (ex: fever, chills, pain, tachycardia, hypotension), laboratory (leukocytosis) and radiologic findings (thick walled, rim-enhancing collection with gas bubbles or air-fluid levels) compatible with an abscess that requires image-guided percutaneous drainage
* Abscess cavity diameters will be less than or equal to 8 cm. However, abscess can be complex or loculated
* Approval by the primary care team to pursue PDT and discuss enrollment with the patient

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergy to contrast media, narcotics, sedatives, atropine or eggs
* Necrotic tissue that requires surgical debridement
* Severely compromised cardiopulmonary function or hemodynamic instability
* Thrombocytopenia (<50,000/mm3)
* Uncorrectable coagulopathy
* Poor kidney function (serum creatinine >3mg/dl)
* Lack of a safe pathway to the abscess or fluid collection
* Unable or unwilling to understand or to provide informed consent
* Unable or unwilling to undergo study procedures
* Patient unable to cooperate with, or to be positioned for the procedure
* Unable to comply with necessary follow up
* Abscesses greater than 8 cm in diameter, multiple separate abscesses in different locations, and abscesses not amenable to safe percutaneous image-guided drainage.
* Patient is currently taking serotonergic psychiatric medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Number of study-related serious adverse events | Up to 14 days post-procedure
Number of patients with study-related unanticipated adverse events | Up to 14 days post-procedure
Evidence of fat embolism | Within 4 hours of Intralipid administration
  Presentation of symptoms, including tachycardia, tachypnea, respiratory failure, decline in hematocrit, thrombocytopenia, and alteration of mental status in patient, will be deemed an unsafe outcome
Methylene blue escape during procedure with evidence of adverse reaction | Within 4 hours of methylene blue administration
  If greater than 3 mg/kg of methylene blue escapes from the abscess (i.e. is not recovered), subject will be placed under observation for 4 hours. During this time, methylene blue related adverse reactions will be assessed. Presence of any of these adverse reactions during the observation period will be considered a safety failure.
Disruption of the abscess wall and damage to surrounding tissue | Up to 14 days post-procedure
  CT imaging post-procedure will be compared to pre-drainage CT imaging for evidence of disruption of the abscess wall and damage to surrounding tissue
Need for surgery to remove a broken optical fiber fragment | Within 1 hour of the study procedure
  If an optical fiber breaks within the patient and surgery is required to retrieve the fragment, this will be deemed an unsafe outcome
Number of patients with technically successful procedure | Within one hour of the trial procedure
  Technical success includes successful image-guided placement of drainage catheter into the abscess, administration of methylene blue and Intralipid, placement of the optical fiber, laser irradiation, and successful removal of the entire optical fiber

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Baran, PhD, Principal Investigator — University of Rochester; Ashwani K Sharma, MD, Principal Investigator — University of Rochester; Laurie Christensen, BS, Study Director — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Haidaris CG, Foster TH, Waldman DL, Mathes EJ, McNamara J, Curran T. Effective photodynamic therapy against microbial populations in human deep tissue abscess aspirates. Lasers Surg Med. 2013 Oct;45(8):509-16. doi: 10.1002/lsm.22171. Epub 2013 Aug 29. PMID 23996629
- [Derived] Baran TM, Bass DA, Christensen L, Longbine E, Favella MD, Foster TH, Sharma AK. Safety and Feasibility of Photodynamic Therapy for Percutaneous Image-guided Abdominopelvic Abscess Drainage: Phase 1 Trial. Radiology. 2024 Mar;310(3):e232667. doi: 10.1148/radiol.232667. PMID 38501946
- [Derived] Hannan MN, Sharma AK, Baran TM. First in human measurements of abscess cavity optical properties and methylene blue uptake prior to photodynamic therapy by in vivo diffuse reflectance spectroscopy. J Biomed Opt. 2024 Feb;29(2):027002. doi: 10.1117/1.JBO.29.2.027002. Epub 2024 Feb 27. PMID 38414658
- [Derived] Li Z, Hannan MN, Sharma AK, Baran TM. Treatment planning for photodynamic therapy of abscess cavities using patient-specific optical properties measured prior to illumination. Phys Med Biol. 2024 Feb 28;69(5):055031. doi: 10.1088/1361-6560/ad2635. PMID 38316055
- [Derived] Li Z, Hannan MN, Sharma AK, Baran TM. Treatment planning for photodynamic therapy of abscess cavities using patient-specific optical properties measured prior to illumination. medRxiv [Preprint]. 2023 Nov 6:2023.10.23.23297420. doi: 10.1101/2023.10.23.23297420. PMID 37961683
- [Derived] Baran TM, Sharma AK. Photodynamic Therapy of an Abdominal Abscess at the Time of Percutaneous Drainage. Cardiovasc Intervent Radiol. 2023 Sep;46(9):1292-1294. doi: 10.1007/s00270-023-03504-z. Epub 2023 Jul 18. No abstract available. PMID 37464107